CLINICAL TRIAL: NCT05037708
Title: Effects of Physiotherapy in the Maintenance Phase in the Treatment of Lymphedema After Breast Cancer
Brief Title: Effects of Physiotherapy in the Treatment of Lymphedema After Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vigo (Other)
Collaborators: Asociación Gallega de Linfedema (Unknown)
Responsible Party: Principal Investigator, Eva María Lantarón Caeiro, Principal Investigator, University of Vigo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Fisioterapia en Linfedema
Record Dates: First submitted 2021-07-19; First posted 2021-09-08 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Lymphedema of Upper Limb
Keywords: Lymphedema of Upper Limb; Breast Neoplasms; Physical Therapy Modalities
MeSH Terms: conditions — Breast Neoplasms | interventions — Manual Lymphatic Drainage

STUDY DESIGN:
Intervention Model Description: Therefore, a randomized, blinded, crossover clinical trial is suggested to assess the effect of an intensive physiotherapy intervention on the treatment of lymphedema in its maintenance phase, in comparison with a control group without physiotherapy treatment.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Group 1 receives treatment A for 4 weeks. Afterwards, a period of washing or bleaching should be allowed in order to be sure that the effects of the intervention have disappeared. This period will last 2 months during which the usual treatment for LGA patients will be carried out, which consists of 2 monthly physiotherapy sessions, in this way it is intended that the subjects are in the initial state (as before the start of the first intervention). After this washout period, treatment B was applied to group 1.
  Interventions: Procedure: Manual lymphatic drainage
- Group 2 (Active Comparator): Group 2 receives treatment B for 4 weeks. Afterwards, a period of washing or bleaching should be allowed in order to be sure that the effects of the intervention have disappeared. This period will last 2 months during which the usual treatment for LGA patients will be carried out, which consists of 2 monthly physiotherapy sessions, in this way it is intended that the subjects are in the initial state (as before the start of the first intervention). After this washout period, treatment A was applied to group 2 .
  Interventions: Procedure: Manual lymphatic drainage

INTERVENTIONS:
Procedure: Manual lymphatic drainage — Subjects are randomly assigned to group 1. Group 1 receives treatment A* for 4 weeks.
  Afterwards, a period of washing or bleaching should be allowed in order to be sure that the effects of the intervention have disappeared. This period will last 2 months during which the usual treatment for LGA patients will be carried out, which consists of 2 monthly physiotherapy sessions, in this way it is intended that the subjects are in the initial state (as before the start of the first intervention). After this washout period, treatment B** was applied to group 1 for 4 weeks.
  *Treatment A consists of manual lymphatic drainage.
  **Treatment B consists of no treatment
  Arms: Group 1
Procedure: Manual lymphatic drainage — Subjects are randomly assigned to group 2. Group 2 receives treatment B** for 4 weeks.
  Afterwards, a period of washing or bleaching should be allowed in order to be sure that the effects of the intervention have disappeared. This period will last 2 months during which the usual treatment for LGA patients will be carried out, which consists of 2 monthly physiotherapy sessions, in this way it is intended that the subjects are in the initial state (as before the start of the first intervention). After this washout period, treatment A* was applied to group 2 for 4 weeks.
  *Treatment A consists of manual lymphatic drainage.
  **Treatment B consists of no treatment
  Arms: Group 2

SUMMARY:
Lymphedema related to breast cancer is one of the main complications after breast cancer treatment. Manual lymphatic drainage appears as a technique which could be applied in the treatment of lymphedema along with other techniques. The aim of this study is to analyze the effects of a physiotherapy program based on manual lymphatic drainage on the treatment of lymphedema after breast cancer, during the stabilization or maintenance phase of complex decongestant therapy. Therefore, a randomized, blinded, crossover clinical trial is suggested to assess the effect of an intensive physiotherapy intervention on the treatment of lymphedema in its maintenance phase, in comparison with a control group without physiotherapy treatment. The cytometry, displaced water volume, thickness of the lymphedema with ultrasound, dynamometry and sensation of heaviness, pain and tension of the upper limb will be evaluated.

DETAILED DESCRIPTION:
Complex decongestant therapy is a set of techniques which seek the treatment of lymphedema in a conservative way as described in the recent international consensus of the International Lymphology Society, published in 2020. Complex decongestant therapy in a first phase aims to reduce cutaneous edema and in a second phase it aims to preserve and optimize the results obtained.

The first phase consists of skin care, manual lymphatic drainage, muscle pumping exercises, and compression techniques, typically applied with multilayer bandages. The second phase consists of compression with low elasticity, skin care exercises, and repeated manual lymphatic drainage as needed.

The frequency and intensity of components of complex decongestant therapy in phase I and II should depend on the clinical findings of edema and the stage of lymphedema and could be adapted to clinical changes. Note that phase II or stabilization represents long-term therapy over many years and in the case of deterioration of edema, phase I of complex decongestant therapy may need to be repeated.

In recent years, there is debate about the efficacy of manual lymphatic drainage. Sometimes it is not prescribed, being replaced by the recommendation of a self-massage. Furthermore, complex decongestant therapy was suggested to be time consuming, expensive and difficult to tolerate, and does not improve lymphatic function.

In contrast, researchers such as Müller et al., in 2018, state that it is a well-tolerated and safe treatment technique, demonstrating benefits in reducing edema. Other research has also shown that manual lymphatic drainage is effective both on a preventive level and as a postoperative rehabilitation treatment, having optimal results when combined with the other elements of complex decongestant therapy.

A recent systematic review published in 2020 highlights the need of more experimental studies on the effectiveness of manual lymphatic drainage on lymphedema. Thus, the

purpose of this study is to analyze the effects of a physiotherapy program based on manual lymphatic drainage in the treatment of lymphedema after breast cancer, during the stabilization or maintenance phase of complex decongestant therapy. Therefore, a double-blind crossover clinical trial is proposed.

ELIGIBILITY:
Inclusion Criteria:

* Women included in the lymphedema treatment maintenance program through the Galician Lymphedema Association
* Women with secondary unilateral lymphedema after breast cancer

Exclusion Criteria:

* Women undergoing chemotherapy or radiotherapy treatment.
* Severe systemic or neurological disease

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-10-27 (Actual)

PRIMARY OUTCOMES:
circometry | 1 day
  measurement of upper limb perimeters
circometry | 1 month
  measurement of upper limb perimeters
circometry | 3 month
  measurement of upper limb perimeters
circometry | 4 month
  measurement of upper limb perimeters
Volumetry by water displacement | 1 day
  weight of water extravasated when introducing the upper limb into a container with water
Volumetry by water displacement | 1 month
  weight of water extravasated when introducing the upper limb into a container with water
Volumetry by water displacement | 3 month
  weight of water extravasated when introducing the upper limb into a container with water
Volumetry by water displacement | 4 month
  weight of water extravasated when introducing the upper limb into a container with water
Measurement of edema thickness by ultrasound | 1 day
  measurement of subcutaneous tissue thickness
Measurement of edema thickness by ultrasound | 1 month
  measurement of subcutaneous tissue thickness
Measurement of edema thickness by ultrasound | 3 month
  measurement of subcutaneous tissue thickness
Measurement of edema thickness by ultrasound | 4 month
  measurement of subcutaneous tissue thickness

SECONDARY OUTCOMES:
Assessment of the sensation of heaviness | 1 day
  Visual analogic scale
Assessment of the sensation of heaviness | 1 month
  Visual analogic scale
Assessment of the sensation of heaviness | 3 month
  Visual analogic scale
Assessment of the sensation of heaviness | 4 month
  Visual analogic scale
Assessment of the sensation of pain | 1 day
  Visual analogic scale
Assessment of the sensation of pain | 1 month
  Visual analogic scale
Assessment of the sensation of pain | 3 month
  Visual analogic scale
Assessment of the sensation of pain | 4 month
  Visual analogic scale
Assessment of the sensation of tension in the upper limb | 1 day
  Visual analogic scale
Assessment of the sensation of tension in the upper limb | 1 month
  Visual analogic scale
Assessment of the sensation of tension in the upper limb | 3 month
  Visual analogic scale
Assessment of the sensation of tension in the upper limb | 4 month
  Visual analogic scale
dynamometry | 1 day
  Assessment of muscle grip strength by dynamometry
dynamometry | 1 month
  Assessment of muscle grip strength by dynamometry
dynamometry | 3 month
  Assessment of muscle grip strength by dynamometry
dynamometry | 4 month
  Assessment of muscle grip strength by dynamometry

CONTACTS AND LOCATIONS:
Overall Officials: Eva M Lantarón_Caeiro, Dra, Principal Investigator — Physiotherapy Group (FS1) - Faculty of Physiotherapy -University of Vigo
Locations (1):
- Faculty of Physiotherapy, Pontevedra, Spain

IPD SHARING:
Plan to Share IPD: No